CLINICAL TRIAL: NCT03825679
Title: Association Between the Composition of the Bacterial Flora of Thrombi and the Etiological Origin of Cerebral Infarctions Treated With Thrombectomy
Brief Title: Association Between the Composition of the Bacterial Flora of Thrombi and the Etiological Origin of Cerebral Infarction Treated With Thrombectomy
Acronym: Bacillus
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BEJOT 2018
Record Dates: First submitted 2019-01-25; First posted 2019-01-31 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Patient With Symptomatic Cerebral Infarction; Patient Who Has Had a Mechanical Thrombectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral infarction is a major health problem. The two most common causes are atherosclerosis (30 to 35%) and cardio-embolic origin (35 to 40%). However, in 25% of cases the cause is undetermined, known as cryptogenic stroke or stroke of undetermined origin. Paroxysmal Atrial Fibrillation appears to cause a significant proportion of these cryptogenic cerebral infarctions. One of the major challenges in the management of cerebral infarctions is the prevention of recurrence. If the cause is atheromatous, treatment is based on platelet antiaggregants and the correction of cardiovascular risk factors. If the cause is atrial fibrillation, the treatment of choice is anticoagulation therapy. Cryptogenic strokes are managed with antiplatelet therapy. In past studies, the thrombi responsible for cerebral infarctions have been analyzed anatomopathologically to see if the composition of the thrombi could help identify the cause of the cerebral infarction. These studies have proved to be contradictory. The composition of the bacterial flora of cerebral infarct thrombi has not yet been studied, apart from some limited data on septic emboli. In myocardial infarction, the cause of which is almost exclusively atheromatous, bacteria of the periodontal flora have been detected in thrombi of ST-segment elevation infarctions. The causes of cerebral infarction are multiple. The hypotheses explored in this study are that there are differences in the composition of the bacterial flora of the thrombus depending on whether the cause is atheromatous or cardio-embolic and that the study of the composition of the thrombus could be used to identify the cardio-embolic cause in patients with cryptogenic cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent (or a close relative or legal representative if the patient is unable to give consent)
* Patient with a symptomatic cerebral infarction defined according to WHO criteria, who has had a mechanical thrombectomy and was hospitalized at the Neurovascular Intensive Care Unit of the Dijon University Hospital.
* 18 years or older

Exclusion Criteria:

* Person not affiliated to national health insurance
* Person under legal protection (curatorship, guardianship)
* Person under court order
* Pregnant or breastfeeding
* Patient who refuses to participate in the study
* Patient (or family member) not reachable by telephone during follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized at the Neurovascular Intensive Care Unit at the Dijon University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2020-01-04 (Actual)

PRIMARY OUTCOMES:
Bacterial composition of thrombi from cerebral infarctions of atheromatous origin and thrombi of cardio-embolic origin | Through study completion, an average of 2 years
  Comparison of the bacterial composition of thrombi from cerebral infarctions of atheromatous origin and thrombi of cardio-embolic origin.
Bacterial composition of cardio-embolic thrombi | Through study completion, an average of 2 years
  Comparison of the bacterial composition of thrombi from cerebral infarctions of atheromatous origin and thrombi of cardio-embolic origin.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France